CLINICAL TRIAL: NCT00333307
Title: A Phase I Randomized, Double-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety of Recombinant Human Relaxin (rhRlx) in Subjects With Preeclampsia
Brief Title: Evaluation of the Safety of Relaxin in Preeclampsia
Status: Suspended | Phase: Phase 1 | Type: Interventional
Sponsor: Corthera, Inc.(formerly BAS Medical, Inc.), a member of the Novartis group of companies (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RLX.PE.001
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Pre-Eclampsia
Keywords: relaxin; preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

INTERVENTIONS:
Drug: recombinant human relaxin

SUMMARY:
The purpose of this study is to determine whether different doses of recombinant human relaxin is safe when given to women with severe preeclampsia

DETAILED DESCRIPTION:
The effects of relaxin may be beneficial in the treatment of women with preeclampsia. This study will preliminarily evaluate the maternal, fetal and neonatal safety and tolerability of an IV infusion of relaxin compared with placebo given to women with severe preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of preeclampsia
* Hospital admission for expectant management

Exclusion Criteria:

* Eclampsia or history of seizures
* Vaginal bleeding
* Multifetal gestation
* Requirement for immediate delivery

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
maternal adverse experiences
fetal adverse experiences
neonatal adverse experiences

SECONDARY OUTCOMES:
preeclampsia assessments
vital signs
physical examinations
clinical laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Sam Teichman, MD, Study Director — Corthera, Inc.(formerly BAS Medical, Inc.), a member of the Novartis group of companies
Locations (2):
- United States (2):
  - Central Baptist Hospital, Lexington, Kentucky
  - University of Cincinnati, Cincinnati, Ohio